CLINICAL TRIAL: NCT05118893
Title: Randomized Ablation-based Atrial Fibrillation Rhythm-control Versus Rate-control Trial in Patients With Heart Failure and High-burden Atrial Fibrillation Extend
Brief Title: Randomized Ablation-based AF Rhythm-control Versus Rate-control in Patients With HF and High-burden AF Extend
Acronym: RAFT-AF Extend
Status: Completed | Type: Observational
Sponsor: Anthony Tang (Other)
Responsible Party: Sponsor-Investigator, Anthony Tang, Professor of Medicine, Western University, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: V15Sep21
Record Dates: First submitted 2021-10-06; First posted 2021-11-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Heart Failure
Keywords: atrial fibrillation; heart failure; long-term follow up
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ablation-based rhythm-control: Ablation-based rhythm-control consisted of pulmonary vein isolation in paroxysmal atrial fibrillation, and additional ablation for persistent atrial fibrillation
- Rate-control: Rate-control included AV-nodal blocking agents and AV node ablation with permanent pacing

SUMMARY:
This is an extended follow up study of the original RAFT-AF Study. The RAFT-AF study was a multi-centre randomized controlled trial with a prospective randomized open blinded endpoint trial (PROBE) design. Patients were randomized to either catheter ablation-based rhythm control of AF as compared to rate control of AF

DETAILED DESCRIPTION:
The RAFT-AF Extend Trial is a continued follow up of patients enrolled in the original RAFT-AF Study (ClinicalTrials.gov, NCT01420393), which evaluated whether ablation-based rhythm-control compared to rate-control improves clinical outcomes in patients with heart failure and atrial fibrillation. It was a randomised, open-label clinical trial, with blinded endpoint adjudication, conducted in 21 institutions in four countries. Patients with atrial fibrillation, New York Heart Association class II-III heart failure, and elevated NT-proBNP were included. Patients were randomized (1:1) to ablation-based rhythm-control or rate-control, stratified by left ventricular ejection fraction (≤45% and >45%). Ablation-based rhythm-control consisted of pulmonary vein isolation in paroxysmal atrial fibrillation, and additional ablation for persistent atrial fibrillation. Rate-control included AV-nodal blocking agents and AV node ablation with permanent pacing. The primary outcome was a composite of mortality and heart failure events, with a minimum follow up of two years. Secondary outcomes included left ventricular ejection fraction, quality of life, six-minute walk test and NT-proBNP. The primary analysis was intention-to-treat. From December 1, 2011, to January 20, 2018, 411 patients were randomised to ablation-based rhythm-control (n=214) or rate-control (n=197). The primary outcome occurred in 50 (23·4%) patients in the ablation-based rhythm-control group and 64 (32·5%) patients in the rate-control group (hazard ratio 0·71 95% CI (0·49, 1·03), p=0·066). Quality of life, six-minute walk distance, left ventricular ejection fraction, and NT-proBNP demonstrated greater improvements in the ablation-based rhythm-control group.

In patients with high burden atrial fibrillation and heart failure, there was no statistically significant reduction of all-cause mortality or heart failure events with ablation-based rhythm-control versus rate-control. With the hazard ratio equivalent to the minimal clinically important difference and the result near statistical significance, there is a probable clinically important benefit of ablation-based rhythm-control over rate-control.

This RAFT-AF Extend study is to extend follow up in RAFT-AF patients for an additional 24 months in order to have sufficient power to definitely determine if ablation-based rhythm control of atrial fibrillation is superior to rate control for the reduction of the primary outcome of all-cause mortality or heart failure event in patient with atrial fibrillation and heart failure.

ELIGIBILITY:
Inclusion Criteria:

All patients previously enrolled and randomized in the RAFT-AF Study that are eligible to enroll

Exclusion Criteria:

* Did not participate in the original RAFT-AF Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients enrolled in the original RAFT-AF Study
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Composite of mortality and Heart Failure Events | 24 months
  Death or HF Event ( admit > 24 hrs or urgent out patient or ER visit for IV diuretics)

SECONDARY OUTCOMES:
all-cause mortality | 24 months
  Death
Heart Failure Events | 24 months
  HF Event ( admit > 24 hrs or urgent out patient or ER visit for IV diuretics)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Tang, Principal Investigator — London Health Sciences Research Institute
Locations (11):
- Canada (11):
  - Libin Cardiovascular Institute, Calgary, Alberta
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - Queen Elizabeth II Health Science, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Science Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUS Le Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec